CLINICAL TRIAL: NCT06840938
Title: Effects of Physiological Manipulation and Surface Electrical Stimulation Towards Safe Swallowing in Post Stroke Dysphagia Patients
Brief Title: Physiological Manipulation and Surface Electrical Stimulation in Post Stroke Dysphagia Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Riphah International University (Other)
Collaborators: Mayo Hospital Lahore (Other)
Responsible Party: Principal Investigator, Nazia Mumtaz, Professor, Head Of Department Speech Language Pathology, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nazia Mumtaz; Arshad Mehmood Naz (Other: Mayo Hospital Lahore)
Record Dates: First submitted 2025-01-17; First posted 2025-02-21 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Dysphagia Following Cerebrovascular Accident
Keywords: Physiological Manipulation; Electrical Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): physiological (maneuvers and positioning)
  Interventions: Behavioral: physiological maneuver
- Group B (Experimental): surface electrical stimulation
  Interventions: Device: Surface Electrical Stimulation
- Group C (Active Comparator): combination of physiological and surface electrical stimulation
  Interventions: Combination Product: Surface Electrical Stimulation

INTERVENTIONS:
Behavioral: physiological maneuver — Group A will be subjected to physiological and postural trainings (traditional)
  Arms: Group A
Device: Surface Electrical Stimulation — Group B will be subjected to Surface Electrical Stimulation through the use of electrodes and stimulators.
  Arms: Group B
Combination Product: Surface Electrical Stimulation — Group C will be subjected to both physiological and Surface Electrical Stimulation supports.
  Arms: Group C

SUMMARY:
Dysphagia is common diagnosed problem after stroke in geriatric population. Digestive system is one of the key systems of human body in which the ingested food is broken down, softened and manipulated in the form of a bolus before actual swallowing. Later however the bolus reaches the stomach where the further disintegration of food is ascertained before it is sent out to intestines where actual absorption of nutrients takes place. A highly active neurological and physiological status ensures a safe travel of food from oral cavity to stomach which otherwise may pose risk of aspiration. Such debilitating conditions are more scientifically known as dysphagia and may present themselves in the form of challenges at oral, pharyngeal and esophageal levels. Although oropharyngeal phase is considered as the key factor leading to aspiration, severe dietary, nutritional and pulmonary challenges may also result. The rehabilitation and efficacy of treatment is seriously linked to an immaculate diagnosis and therapy options available. This study is dedicated to find the effects of present day options including physiological manipulation and surface electrical stimulations for patients who have had developed dysphagia as a result of stroke. It further aims to find the prevailing trends and options available to SLP's rendering services for dysphagia management.

The study is conceived utilizing a mixed method approach whereby both qualitative and quantitative designs will be benefitted. One population of the study comprise stroke patients in the age range of 30-65 years diagnosed to have dysphagia and seeking help at public and private hospitals in Lahore district. A purposive sampling technique will be utilized to select the sample. The sample will be divided into three experimental groups and will be subjected to different treatment options. The treatment will continue for a period of 12 weeks and later will be evaluated in pre-post comparisons in terms of severity of dysphagia. Data will be interpreted in terms of percentages, frequencies and means etc., etc. An inferential statistical comparison (one way Anova) will be conducted to find any significant difference in the treatment groups.

Another population of the study will comprise speech language professionals rendering services to dysphagic patients, conveniently sampled and interviewed. The qualitative analysis will yield information about present day options and preferences among SLP's for respective audience.

ELIGIBILITY:
Inclusion Criteria:

* post stroke Dysphagia patients will be included.

Exclusion Criteria:

* Any other co-morbid condition (Parkinson disease, Alzheimer disease) will be excluded.
* Drug intake, History of Alcohol & Smoking will be excluded.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-05 (Estimated)

PRIMARY OUTCOMES:
Severity of dysphagia | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided